CLINICAL TRIAL: NCT01183260
Title: Evaluation of the Trabecular Metal™ Acetabular Revision Cup Using Dual-Energy X-ray Absorptiometry (DEXA)
Brief Title: Evaluation of the Trabecular Metal™ Revision Hip Cup Using Bone Mineral Density (DEXA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Wael Barsoum, MD, Chairman of Surgical Operations, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZIMM1007WB; 09-859 (Other: CCF IRB)
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Revision, Joint
Keywords: revision total hip arthroplasty; bone mineral density; trabecular metal; DEXA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trabecular Metal Revision Cup (Experimental): Patients randomized to this arm will receive a trabecular metal revision component which does not have a titanium inner surface and requires a cemented highly crosslinked polyethylene liner.
  Interventions: Device: Trabecular Metal Revision Cup
- Trabecular Metal Modular Cup (Active Comparator): Patients randomized to this arm will receive a trabecular metal modular component which has a titanium inner surface and requires a non-cemented highly crosslinked polyethylene liner.
  Interventions: Device: Trabecular Metal Modular Cup

INTERVENTIONS:
Device: Trabecular Metal Revision Cup — Revision of the acetabular cup
  Arms: Trabecular Metal Revision Cup
Device: Trabecular Metal Modular Cup — Revision of the acetabular cup
  Arms: Trabecular Metal Modular Cup

SUMMARY:
In 1997, the FDA approved the use of Trabecular Metal™ (Zimmer, Trabecular Metal Technology, Inc., Parsippany, NJ) for acetabular cups, a porous tantalum structural biomaterial that was developed to address the limitations of other implant materials, with the potential to improve implant fixation.

Porous tantalum (80% porosity) offers potentially greater ingrowth and bone graft incorporation, believed to be restricted by the low porosity of other commonly used implants (30%). Additionally, the low modulus of elasticity property (3 MPa) of porous tantalum provides more normal physiological loading conditions which theoretically reduce stress shielding and resultant bone loss surrounding the implant. These properties are much desired advantages for implants used in cementless THA.

Various porous tantalum implants have shown favorable clinical results. Unger et al. reported excellent bone graft incorporation of the acetabular component based on serial radiograph data at a minimum 1-year follow-up.

Dual-energy X-ray absorptiometry (DEXA) is a well-established method for detecting periprosthetic bone mass changes around the femoral and acetabular THA components.

The primary objective of this study is to quantify and compare periprosthetic bone mineral density (BMD) changes in THA revision patients receiving Trabecular Metal™ and metal-backed acetabular components, measured using DEXA scanning techniques. Additionally, this study will analyze and compare clinical outcomes of these patients, based on SF-12v2 and HOOS.

DETAILED DESCRIPTION:
none provided.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 85 years
* Sex: Both male and female will be included. The male-to-female ratio will depend upon the patient population.
* Stable Health: At the time of surgery based on physical examination and medical history.
* Patient is a revision total hip recipient, which requires a metal-backed hemispherical cup.
* Patient or patient's legal representative has signed the Informed Consent form. The patient is capable of making informed decisions regarding his/her healthcare.

Exclusion Criteria:

* Patients undergoing bilateral surgery or had prior hip arthroplasty on contralateral side less than 6 months from date of surgery.
* Patients who do not plan to return to a Cleveland Clinic surgeon for follow-up visits (i.e. out of state/country patients who may choose to follow-up with a different surgeon).
* Patients with history of radiation therapy.
* Patients with known diagnosis of Brooker grade 3 or 4 HO (heterotopic ossification) in the hip joint region.
* Patients with known diagnosis of renal disease.
* Patients with known diagnosis of osteoporosis.
* Patients with history of steroid use in the hip joint region.
* Patients that have had a previous lumbar fusion.
* Patients whose surgical reconstruction required a pelvic cage or plate.
* Patient was a poor compliance risk - treated for ethanol or drug abuse, physical or mental handicap, etc.
* Any female of childbearing potential who is pregnant or is planning on becoming pregnant during the study period (~2 years postoperative).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-08; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wael K Barsoum, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 2010 - 2014
Groups:
- Zimmer Trabecular Metal Acetabular Cup: Zimmer Trabecular Metal Revision Cup: Revision of the acetabular cup
- Zimmer Modular Cup: Zimmer Modular Cup: Revision of the acetabular cup
Period: Overall Study
Arm/Group | Zimmer Trabecular Metal Acetabular Cup | Zimmer Modular Cup
Started | 14 | 11
Completed | 10 | 9
Not Completed | 4 | 2
Not completed — Intraop screen failure | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Revised within 30 days | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zimmer Trabecular Metal Acetabular Cup | Zimmer Modular Cup | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.60 (11.40) | 61.11 (9.74) | 59.79 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 19
Operative Side: Left, Right [Count of Participants; unit: Participants]
  Left | 5 | 5 | 10
  Right | 5 | 4 | 9
BMI (kg/m^2), Continuous [Mean (Standard Deviation); unit: kg/m^2] | 30.14 (6.07) | 30.49 (7.56) | 30.31 (6.44)

OUTCOME MEASURES:

1. Primary Outcome: Periprosthetic Bone Mineral Density (BMD) of Hip
Description: Quantify and compare periprosthetic bone mineral density (BMD) changes in THA revision patients receiving Trabecular Metal™ and metal-backed acetabular components, measured using DEXA scanning techniques. Region 1 forms the superior-lateral region, Region 2 forms the superior-medial region, and Region 3 forms the inferior-medial region around the acetabular component. For each region, the mean change in BMD was calculated using the following equation described by Wilkinson et al (J Bone Joint Surg Br., 2001): mean percent change in BMD = (BMD1-BMD2) x 2 x 100 / (BMD1 + BMD2). These regions were patient specific and remained the same each time the patient was scanned.
Time Frame: 2 years postoperative; measured at 3 months (baseline), 6 months, 1 year, 2 year postoperative
Population: By Year 2, there were 3 patients lost to follow-up in the Revision Cup group and 3 patients lost to follow-up in the Modular Cup group:
  We were unable to contact 1 patient from each group in order to schedule follow-up The remaining patients were withdrawn because they were feeling fine and declined to return for follow-up at that time
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Zimmer Trabecular Metal Acetabular Cup | Zimmer Modular Cup
Number analyzed (Participants) | 10 | 9
g/cm^2
  3 Month - Region 1 | 1.63 (0.42) | 1.64 (0.38)
  3 Month - Region 2 | 1.85 (0.34) | 1.64 (0.31)
  3 Month - Region 3 | 1.27 (0.33) | 0.92 (0.31)
  3 Month - Lumbar Spine (L1-L4) | 1.29 (0.15) | 1.21 (0.18)
  6 Month - Region 1: number analyzed (Participants) | 9 | 9
  6 Month - Region 1 | 1.61 (0.18) | 1.82 (0.28)
  6 Month - Region 2: number analyzed (Participants) | 9 | 9
  6 Month - Region 2 | 1.75 (0.31) | 1.76 (0.33)
  6 Month - Region 3: number analyzed (Participants) | 9 | 9
  6 Month - Region 3 | 1.22 (0.30) | 0.94 (0.30)
  6 Month - Lumbar Spine (L1-L4): number analyzed (Participants) | 9 | 9
  6 Month - Lumbar Spine (L1-L4) | 1.29 (0.17) | 1.22 (0.16)
  1 Year - Region 1: number analyzed (Participants) | 8 | 9
  1 Year - Region 1 | 1.64 (0.17) | 1.84 (0.34)
  1 Year - Region 2: number analyzed (Participants) | 8 | 9
  1 Year - Region 2 | 1.82 (0.28) | 1.72 (0.41)
  1 Year - Region 3: number analyzed (Participants) | 8 | 9
  1 Year - Region 3 | 1.23 (0.14) | 1.22 (0.16)
  1 Year - Lumbar Spine (L1-L4): number analyzed (Participants) | 8 | 9
  1 Year - Lumbar Spine (L1-L4) | 1.26 (0.14) | 1.22 (0.16)
  2 Year - Region 1: number analyzed (Participants) | 7 | 6
  2 Year - Region 1 | 1.75 (0.23) | 1.93 (0.45)
  2 Year - Region 2: number analyzed (Participants) | 7 | 6
  2 Year - Region 2 | 1.76 (0.24) | 1.83 (0.71)
  2 Year - Region 3: number analyzed (Participants) | 7 | 6
  2 Year - Region 3 | 1.19 (0.24) | 1.00 (0.36)
  2 Year - Lumbar Spine (L1-L4): number analyzed (Participants) | 7 | 6
  2 Year - Lumbar Spine (L1-L4) | 1.26 (0.14) | 1.15 (0.14)

2. Secondary Outcome: Functional and General Health Outcome Assessments
Description: Analyze and compare functional and general health outcomes of these patients, based on Hip disability and Osteoarthritis Outcomes Score (HOOS) and 12-item Short Form Health Survey (SF-12v2). All subscale scores are calculated independently and range from 0 to 100, where 100 indicates no problems:
  * SF-12 Physical Component Summary Subscale (SF12 PCS) assesses physical function, bodily pain, and general health.
  * SF-12 Mental Component Summary Subscale (SF12 MCS) assesses emotional and mental health.
  * HOOS Pain assesses pain in the hip
  * HOOS Symptoms assesses symptoms such as stiffness in the hip
  * HOOS activities of daily living (HOOS ADL) assesses physical function while performing common daily activities (walking, sitting, standing, etc.)
  * HOOS sport and recreation (HOOS Sports/Rec) assesses physical function while performing higher-level activities (running, squatting, etc.)
  * HOOS hip-related quality of life (HOOS QOL) assesses how much the hip impacts life
Time Frame: 2 years postoperative; measured preoperatively and 3 months, 6 months, 1 year, 2 year postoperative
Population: By Year 2, there were 3 patients lost to follow-up in the Revision Cup group and 3 patients lost to follow-up in the Modular Cup group:
  We were unable to contact 1 patient from each group in order to schedule follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zimmer Trabecular Metal Acetabular Cup | Zimmer Modular Cup
Number analyzed (Participants) | 10 | 9
units on a scale
  Preop SF12 PCS | 32.25 (5.86) | 38.57 (12.07)
  Preop SF12 MCS | 55.29 (8.07) | 47.62 (10.39)
  3 Month SF12 PCS | 32.25 (8.38) | 38.57 (11.63)
  3 Month SF12 MCS | 51.78 (8.10) | 51.09 (9.45)
  6 Month SF12 PCS: number analyzed (Participants) | 9 | 9
  6 Month SF12 PCS | 32.14 (7.22) | 40.12 (13.00)
  6 Month SF12 MCS: number analyzed (Participants) | 9 | 9
  6 Month SF12 MCS | 50.51 (11.53) | 52.83 (7.70)
  1 Year SF12 PCS: number analyzed (Participants) | 8 | 9
  1 Year SF12 PCS | 31.04 (12.54) | 42.84 (16.14)
  1 Year SF12 MCS: number analyzed (Participants) | 8 | 9
  1 Year SF12 MCS | 55.58 (10.18) | 54.04 (8.64)
  2 Year SF12 PCS: number analyzed (Participants) | 7 | 6
  2 Year SF12 PCS | 36.10 (11.39) | 47.05 (13.52)
  2 Year SF12 MCS: number analyzed (Participants) | 7 | 6
  2 Year SF12 MCS | 53.46 (7.93) | 48.66 (11.24)
  Preop HOOS Pain | 50.25 (20.19) | 36.67 (25.19)
  Preop HOOS Symptoms | 46.50 (18.72) | 38.33 (27.95)
  Preop HOOS ADL | 39.48 (8.63) | 32.11 (31.24)
  Preop HOOS Sports/Rec | 8.75 (12.96) | 15.28 (21.40)
  Preop HOOS QOL | 28.89 (31.95) | 27.16 (25.53)
  3 Month HOOS Pain | 61.50 (16.72) | 76.39 (17.37)
  3 Month HOOS Symptoms | 55.50 (19.50) | 66.67 (18.03)
  3 Month HOOS ADL | 52.45 (14.23) | 66.81 (17.09)
  3 Month HOOS Sports/Rec | 21.88 (16.39) | 29.17 (15.80)
  3 Month HOOS QOL | 28.89 (16.73) | 49.38 (30.99)
  6 Month HOOS Pain: number analyzed (Participants) | 9 | 9
  6 Month HOOS Pain | 61.94 (19.07) | 81.94 (14.02)
  6 Month HOOS Symptoms: number analyzed (Participants) | 9 | 9
  6 Month HOOS Symptoms | 58.33 (17.68) | 76.67 (19.04)
  6 Month HOOS ADL: number analyzed (Participants) | 9 | 9
  6 Month HOOS ADL | 55.56 (15.71) | 76.79 (17.15)
  6 Month HOOS Sports/Rec: number analyzed (Participants) | 9 | 9
  6 Month HOOS Sports/Rec | 26.39 (18.00) | 46.13 (29.98)
  6 Month HOOS QOL: number analyzed (Participants) | 9 | 9
  6 Month HOOS QOL | 37.04 (23.57) | 49.38 (37.31)
  1 Year HOOS Pain: number analyzed (Participants) | 8 | 9
  1 Year HOOS Pain | 61.88 (27.57) | 81.67 (12.18)
  1 Year HOOS Symptoms: number analyzed (Participants) | 8 | 9
  1 Year HOOS Symptoms | 63.75 (30.68) | 75.83 (18.03)
  1 Year HOOS ADL: number analyzed (Participants) | 8 | 9
  1 Year HOOS ADL | 56.88 (26.80) | 76.88 (17.77)
  1 Year HOOS Sports/Rec: number analyzed (Participants) | 8 | 9
  1 Year HOOS Sports/Rec | 20.49 (20.68) | 51.49 (19.79)
  1 Year HOOS QOL: number analyzed (Participants) | 8 | 9
  1 Year HOOS QOL | 38.89 (31.98) | 56.79 (37.45)
  2 Year HOOS Pain: number analyzed (Participants) | 7 | 6
  2 Year HOOS Pain | 69.64 (26.71) | 82.92 (24.41)
  2 Year HOOS Symptoms: number analyzed (Participants) | 7 | 6
  2 Year HOOS Symptoms | 65.54 (23.98) | 70.00 (29.83)
  2 Year HOOS ADL: number analyzed (Participants) | 7 | 6
  2 Year HOOS ADL | 66.19 (26.93) | 77.38 (18.65)
  2 Year HOOS Sports/Rec: number analyzed (Participants) | 7 | 6
  2 Year HOOS Sports/Rec | 39.58 (25.43) | 65.83 (20.92)
  2 Year HOOS QOL: number analyzed (Participants) | 7 | 6
  2 Year HOOS QOL | 60.32 (29.99) | 62.96 (24.00)

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Zimmer Trabecular Metal Acetabular Cup | Zimmer Modular Cup
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zimmer Trabecular Metal Acetabular Cup (N=14) | Zimmer Modular Cup (N=11)
Revision surgery due to multiple dislocations (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
A large amount of variability was present in the data leading to reduced statistical power during hypothesis testing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No